CLINICAL TRIAL: NCT05657288
Title: SpO2 Comparison Between Commercial Smartwatch and Medical-grade Pulse Oximeter
Brief Title: SpO2 Comparison Between Commercial Smartwatch and Medical-grade Pulse Oximeter During Hypoxia
Acronym: HYPOWATCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NVT02/2022
Record Dates: First submitted 2022-12-10; First posted 2022-12-20 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Hypoxia; Pulse Oximetry
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Interventional prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypoxia (Experimental): Volunteers sequentially inhale three hypoxic gas mixtures each for 2.5 minute. Every measurement will begin with a two-minute stabilization phase, during which the physiological values of the volunteer will be checked. During the whole experiment, non-invasive SpO2 measurements will be performed on the middle finger and on the wrist of left hand.
  Interventions: Other: Breathing mixtures of O2 and N2 and monitoring SpO2 on finger and left wrist

INTERVENTIONS:
Other: Breathing mixtures of O2 and N2 and monitoring SpO2 on finger and left wrist — Volunteers sequentially inhale three hypoxic gas mixtures each for 2.5 minute. Every measurement will begin with a two-minute stabilization phase, during which the physiological values of the volunteer will be checked. During the whole experiment, non-invasive SpO2 measurements will be performed on the middle finger and on the wrist of left hand.

SUMMARY:
The aim of the project is to experimentally compare SpO2 measured on a wrist by commercial Smartwach and on a finger measured by a medical-grade pulse oximeter in healthy humans during gradual desaturation in the range of 60-100% SpO2 and simultaneously during a step change from the hypoxic phase to the recovery phase (return to physiological values).

DETAILED DESCRIPTION:
The newest models of smartwatches measure peripheral blood oxygen saturation (SpO2) and the technology is rapidly improving. The results of individual studies on the accuracy of SpO2 measurement using smartwatches from different brands are still inconclusive. The study aims to compare the measurement of peripheral blood oxygen saturation using the latest smartwatch with a medical-grade pulse oximeter under the condition of normobaric hypoxia. SpO2 measurements will be taken by hand from the watch and the pulse oximeter simultaneously. The agreement of the measurements of both devices will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Passing the initial examination, which will determine the following data: finger circumference, heart rate, blood pressure, blood oxygen saturation and medical history

Exclusion Criteria:

* pregnancy
* severe cardiovascular conditions
* severe asthma or other severe respiratory conditions
* injury to the upper limbs or hands that could affect the peripheral perfusion
* diabetes
* hypotension or hypertension

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-05-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Is there any difference in measured SpO2 between finger and wrist during induced hypoxia? | 1 hour
  The agreement of SpO2 measurements of both monitoring devices will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Walzel, MSc., Principal Investigator — Czech Technical University
Locations (1):
- Czech Technical University in Prague, Kladno, Czechia

REFERENCES:
- [Background] Rafl J, Bachman TE, Rafl-Huttova V, Walzel S, Rozanek M. Commercial smartwatch with pulse oximeter detects short-time hypoxemia as well as standard medical-grade device: Validation study. Digit Health. 2022 Oct 11;8:20552076221132127. doi: 10.1177/20552076221132127. eCollection 2022 Jan-Dec. PMID 36249475